CLINICAL TRIAL: NCT00127907
Title: Comparison of Epinephrine Associated With Vasopressin vs Epinephrine Alone in the Treatment of Out-of-Hospital Cardiac Arrests
Brief Title: Vasopressin and Epinephrine Versus Epinephrine Alone in Cardiac Arrest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003.329
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-10

CONDITIONS: Cardiac Arrest
Keywords: Out-of-hospital cardiac arrest - Vasopressin - Epinephrine
MeSH Terms: conditions — Heart Arrest | interventions — Epinephrine; Arginine Vasopressin

INTERVENTIONS:
Drug: epinephrine (1 mg/1 mL)
Drug: arginine-vasopressin (40 UI/2 mL)

SUMMARY:
Recent studies have suggested that arginine-vasopressin could be more effective in the treatment of cardiac arrests. The last published study did not outline obvious improvements in the prognosis of all cardiac arrests but pointed out a possible increased survival rate when arginine-vasopressin is associated with epinephrine. The aim of this study is to compare the efficacy of two successive injections of epinephrine (1 mg) with two successive injections of epinephrine associated with arginine-vasopressin (40 UI) in out-of-hospital cardiac arrests occurring in adult patients. The primary endpoint is the survival rate at hospital admission. The inclusion period lasts 18 months and 2416 patients are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital medical cardiac arrest in adult patients.

Exclusion Criteria:

* Traumatic cardiac arrest
* Pregnancy
* Patients younger than 18 years old or older than 85 years old

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2416
Dates: Start 2004-05

PRIMARY OUTCOMES:
Survival at hospital admission

SECONDARY OUTCOMES:
ROSC (Return of spontaneous circulation) Survival at : H24, Day 28, hospital discharge and one year Neurological status at H24 and hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves GUEUGNIAUD, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

REFERENCES:
- [Derived] Gueugniaud PY, David JS, Chanzy E, Hubert H, Dubien PY, Mauriaucourt P, Braganca C, Billeres X, Clotteau-Lambert MP, Fuster P, Thiercelin D, Debaty G, Ricard-Hibon A, Roux P, Espesson C, Querellou E, Ducros L, Ecollan P, Halbout L, Savary D, Guillaumee F, Maupoint R, Capelle P, Bracq C, Dreyfus P, Nouguier P, Gache A, Meurisse C, Boulanger B, Lae C, Metzger J, Raphael V, Beruben A, Wenzel V, Guinhouya C, Vilhelm C, Marret E. Vasopressin and epinephrine vs. epinephrine alone in cardiopulmonary resuscitation. N Engl J Med. 2008 Jul 3;359(1):21-30. doi: 10.1056/NEJMoa0706873. PMID 18596271